CLINICAL TRIAL: NCT00398099
Title: Clinical Evaluation for the Efficacy, Safety, Tolerability & Medical Resource Utilization of Invanz (Ertapenem Sodium) Therapy
Brief Title: To Evaluate the Treatment Effect of an Anti-Infective Agent for Different Kinds of Infections (0826-052)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0826-052; 2006_046
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Infection; Pneumonia; Urinary Tract Infection
MeSH Terms: conditions — Infections; Pneumonia; Urinary Tract Infections | interventions — Ertapenem; Duration of Therapy

INTERVENTIONS:
Drug: MK0826, ertapenem sodium / Duration of Treatment: 14 Days

SUMMARY:
To collect clinical response data with the use of ertapenem in approved indications.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 20 years of age or older
* Patients did not receive any systemic antibiotic before enrollment, or patients with failed clinical response (no improvement on symptoms or laboratory data) through previous antibiotic treatment
* Patients who required therapy prior to identification of cause of infection

Exclusion Criteria:

* Patient has a concomitant infection that may interfere with the evaluation of the response to ertapenem
* Patient has an apache ii > 30.
* Patient has an infection caused by pathogens resistant to ertapenem
* Patients with known allergy to ertapenem or other drugs in the same carbapenem class, beta - lactams, lidocaine or local anesthetics of the amide type
* The patient requires antibiotics other than ertapenem (such as: glycopeptides, macrolides or antifungal agents)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-07; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Signs and symptoms of infection on days 3, 4, 7 and 14 during treatment

SECONDARY OUTCOMES:
Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html